CLINICAL TRIAL: NCT00535808
Title: Effect of Strategy for Blood Pressure Control on Cerebral Oxygen Balance During Aortic Coarctation Repair: a Randomized Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007/270
Record Dates: First submitted 2007-09-25; First posted 2007-09-26 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Cerebral Oxygenation
MeSH Terms: interventions — Nitroprusside; Nitroglycerin; Sevoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Administration of nitroprusside
  Interventions: Drug: nitroprusside
- 2 (Experimental): Administration of nitroglycerine
  Interventions: Drug: nitroglycerine
- 3 (Experimental): Administration of sevoflurane
  Interventions: Drug: sevoflurane

INTERVENTIONS:
Drug: nitroprusside — Administration of nitroprusside
  Arms: 1
Drug: nitroglycerine — Administration of nitroglycerine
  Arms: 2
Drug: sevoflurane — Administration of Sevoflurane
  Arms: 3

SUMMARY:
In a prospective and randomized study protocol, three different blood pressure regulating agents (nitroprusside, nitroglycerine, sevoflurane) will be compared concerning their effect on the cerebral oxygen balance between both hemispheres during aortic coarctation repair. Cerebral and somatic saturation will be monitored non-invasively and continuously via optical sensors applied to the right and left forehead and the somatic regions. Arterial blood pressure, central venous pressure, heart rate and systemic saturation will be recorded continuously. Intermittently, arterial and venous blood gas analysis will be performed at 6 definite time intervals. The study ends at the end of the operation.

ELIGIBILITY:
Inclusion Criteria:

* All neonates and infants
* Aged 0-18 year
* With aortic coarctation requiring surgical correction without the additional use of cardiopulmonary bypass will be included.

Exclusion Criteria:

* All patients with an associated cardiac effect are excluded.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2007-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Cerebral saturation | During operation

CONTACTS AND LOCATIONS:
Overall Officials: Annelies Moerman, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be